CLINICAL TRIAL: NCT03583229
Title: ECP Study: Extracorporeal Photopheresis as Treatment of Cardiac Allograft Vasculopathy After Heart Transplantation and Evaluation of Platelet Function and Aggregation After Heart Transplantation
Brief Title: Coronary Artery Disease After Heart Transplantation
Acronym: ECP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Hans Eiskjær, Professor, DMSc, Aarhus University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECP studiet
Record Dates: First submitted 2018-06-27; First posted 2018-07-11 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease in Transplanted Heart (Diagnosis); Platelet Dysfunction
Keywords: Heart Transplantation; Cardiac Allograft Vasculopathy
MeSH Terms: conditions — Disease | interventions — Aspirin; Photopheresis

STUDY DESIGN:
Intervention Model Description: Patients with antibodies receive 4 ECP-treatments if they have CAV. If patients do not want to receive ECP-treatments, they are allocated to the control group, which do not receive ECP-treatments.
  All patients receive 7 days treatment with aspirin and blood samples are drawn before and after.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aspirin - single arm (Other): 1 tablet of Aspirin 75 mg administered x 1 daily for 7 days.
  Interventions: Drug: Aspirin 75mg
- Extracorporeal photopheresis (Experimental): All patients with HLA antibodies receive 4 ECP-treatments in 2 months.
  Interventions: Drug: Aspirin 75mg; Other: Extracorporeal photopheresis
- Control group (No Intervention): The control group does not receive ECP-treatments, but blood samples are drawn at the same intervals as treatment group and CAG+OCT are also performed at baseline and 12 months follow up as the treatment group.

INTERVENTIONS:
Drug: Aspirin 75mg — 7 days treatment with 75 mg aspirin daily.
  Arms: Aspirin - single arm; Extracorporeal photopheresis
Other: Extracorporeal photopheresis — 4 x ECP treatments in 60 days.
  Arms: Extracorporeal photopheresis

SUMMARY:
This study evaluates coronary artery disease after heart transplantation and its relation to platelet function. Furthermore, we will evaluate extracorporeal photopheresis as treatment of coronary artery disease after heart transplantation.

DETAILED DESCRIPTION:
BACKGROUND

Part one:

Heart transplantation (HTX) is an excellent treatment of end stage heart failure with a mean survival of approximately 15.6 years (1). Long-term survival remains a challenge. With improvement of immunosuppressive therapy, incidences of acute cellular rejection (ACR) have declined, but after the first postoperative year, one of the main causes of death is cardiac allograft vasculopathy (CAV), which is an accelerated form of coronary artery disease (2).

ACR is a well-recognized phenomenon but the diagnosis of antibody-mediated rejection (AMR) has gained acceptance. AMR is associated with greater graft dysfunction, development of CAV and mortality. The diagnosis is based on clinical, histopathologic, immunopathologic and identification of donor-specific antibodies by solid phase assays (3,4). However, AMR is often clinically silent, and the histopathologic and immunopathologic evaluation may be associated with significant inter-observer variation. Identification of donor specific antibodies (DSA) could seem more suitable. In the GRAFT study, we found significantly increased levels of DSA in approximately 25% of HTX patients. They had subclinical reduced graft function, higher previous ACR burden and prevalence of CAV.

Guidelines recommend routinely evaluation of DSA, but the evidence of treating patients with DSA and no pathological findings is poor.

Extracorporeal photopheresis (ECP) inactivates lymphocytes and reduce cellular myocardial infiltration and production of DSA. Although the results for treatment of ACR and AMR appear promising, ECP is limited to a few centers (3,5,6).

The aim of this study is to evaluate the impact of ECP on CAV.

Part two:

The cause of CAV after HTx is unknown. CAV is a diffuse, progressive thickening of the arterial intima that develops in both the epicardial and intramyocardial arteries. Optical coherence tomography (OCT) and virtual histology intravascular ultrasound (IVUS) have revealed multilayered plaques in approximately 50% of patients (7), which likely represent intravascular thrombosis (7,8). Autopsy studies conﬁrm a high prevalence (63-83%) of coronary thrombi (9). Platelets are the cellular mediator of thrombosis, but also play an important role in the immune system. Previous studies indicate that platelets are involved in vascular inflammation and immune cell trafficking in acute graft rejection. Platelet ligand induced binding site-1 (LIBS-1) antibody binding is correlated with CAV progression in HTX patients (10). Hence, platelets may play an important role in CAV progression. Further studies are needed to clarify the relation between platelet function and coronary thrombi, and the effect of aspirin on platelet function in HTX patients.

The aim of this part of the study is to evaluate the relationship between platelet function and the presence of luminal thrombi, and the relation between luminal thrombi and the blood clot formation and degeneration.

Platelet function and blood clot formation:

Ischemic heart disease is caused by atherosclerosis. Rupture of an atherosclerotic plaque causes activation of platelets and the coagulation system, ultimately resulting in a thrombus. Recent reports by IVUS (7) and OCT (8) have revealed high prevalence of complexed layered plaques, which might represent organized thrombus.

Coronary flow velocity reserve:

The coronary flow velocity reserve (CFVR) represents the capacity of the coronary circulation to dilate, following an increase in myocardial metabolic demands. CFVR is defined as the ratio of maximum flow/hyperaemic flow under adenosine infusion to resting blood flow velocity in the epicardial coronary arteries (14).

A CFVR value of 2 discriminates significant from non-significant coronary stenosis.

STUDY DESIGN

Controlled prospective study of all patients with CAV and DSA followed at the Department of Cardiology, AUH, Skejby. Based on our calculation sample size would be 30 patients. A graft age matched group of 30 HTX patients without DSA will be included as controls.

METHODS

Patients are screened for eligibility to be included prior to annual routine examinations and informed consent is obtained. CAG, OCT and advanced echocardiography at rest and during exercise including coronary flow reserve (CFR) measurements at baseline and at 12 months follow-up are performed at Department of Cardiology, Aarhus University Hospital. 34 ml blood will be stored in the biobank. Blood samples before and after 7 days treatment with 75 mg aspirin daily.

If DSA levels >3000 MFI with Luminex analysis, the patient receives ECP treatments at Department of Immunology, Aarhus University Hospital.

Platelet function:

Is evaluated by whole blood platelet aggregometry using Multiplate® Analyzer. This instrument is based on impedance aggregometry, in which the level of platelet aggregation is reflected by changes in impedance between two electrodes. Arachidonic acid (ASPI test), TRAP-6 and adenosine diphosphate (ADP test) are used as agonists to induce platelet aggregation. For verification of aspirin compliance, serum thromboxane B2 levels will be measured.

Platelet turnover parameters are evaluated using automated flow cytometry (Sysmex XN 9000). Platelet count, immature platelet fraction and count, mean platelet volume, platelet distribution width and platelet large-cell-ratio are measured.

Coronary angiography (CAG):

An experienced operator will perform CAG according to routine protocol after HTx. The degree of CAV will be quantified in a blinded fashion according to ISHLT guidelines:

* CAV 0: No stenosis/irregularity
* CAV 1: <70% major branch or <50% left main stem
* CAV 2: >70% major branch or >50% left main stem with normal diastolic graft function
* CAV 3: >70% major branch or >50% left main stem with impaired diastolic graft function.

Optical coherence tomography (OCT):

OCT acquisition is performed in all three major coronary arteries during CAG by use of Terumo Lunawave system as advised by the manufacturer and according to department standard operating procedure. Analysis is performed in a blinded fashion using the QCU-CMS software (Leiden University Medical Center, NL). Quantitative intimal tissue analysis is performed in areas without advanced plaque morphology. All plaques in the acquired segments are characterized and sized according to luminal presentation and mapped for serial assessment. Macrophage infiltration is quantified as a marker of inflammation. Layered complex plaques are defined as a heterogenic signal in intima with a layered structure.

The patients are divided in three groups according to the extent of CAV by complex layered plaques:

* 0 %
* 0-7 %
* >7 %

Transthoracic echocardiography:

The following parameters will be recorded: 2D ejection fraction, regional wall motion score (17 segment model), left ventricular end diastolic (LVEDV) and systolic volume (LVESV), left atrial volume, tissue Doppler study of the mitral annulus and LV strain and strain-rate. Furthermore, diastolic function will be evaluated by early diastolic myocardial velocity, E/A ratio, EdecT, isovolumetric relaxation time (IVRT) and E/e' ratio. Global longitudinal strain (GLS) will be assessed from two-dimensional images of the apical four-chamber, two-chamber, and long-axis view with an optimized frame rate (50-90 frames/sec).

Coronary Flow Reserve (CFR) by tissue Doppler echocardiography:

The distal LAD is localized and the flow velocity is measured with Doppler using a 6 MHz probe at basal conditions and during adenosine infusion (hyperemia) at 140 µg/kg/min.

Exercise Protocol:

We will measure peak oxygen consumption by cardiopulmonary exercise test (CPX). The patients will perform a multistage symptom limited semi supine cycle ergometer exercise test using GE Healthcare eBike L Ergometer (Wauwatosa, WI 53226 U.S.A.). Workload starts at 0 W and increases by 25 W every 3 minutes. Patients will be encouraged to exercise until exhaustion (Borg >18). Brachial blood pressure will be measured at baseline and every 3 minutes until maximum workload is reached.

ECP:

1. Collection of mononuclear cells by apheresis
2. Addition of 8-methoxyspsoralen (8-MOP) to the cells followed by ultraviolet A (UVA) irradiation
3. Reinfusion of the treated cells.

Collection of mononuclear cells will be performed with Spectra Optia using cMNC or MNC software (TerumoBCT, Lakewood, CO, USA) on 2 consecutive days. With MNC, two chamber collections (21 + 4 mL) are performed providing a fixed product volume of 50 mL. With MNC, collection is performed preferably 1 ml/min until a product volume of 75 mL. Hct is measured on a sample taken from the sample tube of the Spectra Optia kit. The product is diluted with 250 ml NaCl to an end volume of 300 ml. The product bag is sterile connected to the illumination bag and 3 mL 8-MOP (Macopharma, Tourcoing, France) is added to the product. Illumination is performed in Macogenic G2 (Macopharma, Tourcoing, France). The Hct before addition of 8-MOP should not exceed 2 %. Documentation and traceability are maintained by using blood bank IT system (Prosang, Databyrån, Stockholm, Sweden) and ISBT128 labeling.

SAMPLE SIZE CALCULATION - PLATELET FUNCTION

>Sample size calculation based on data from healthy volunteers off-aspirin<

The primary outcome is the difference in platelet aggregation between HTx patients with and without CAV and healthy volunteers. No publications report platelet aggregation in HTx patients but from a previous study we know that the mean platelet aggregation in healthy drug-naive individuals is 1004 aggregation units x minute with a standard deviation of 163 aggregation units x minute using arachidonic acid (AA) as agonist (ASPI-test). Choosing a minimal relevant difference of 150 aggregation units x minute, a significance level (two-sided alpha) of 5%, and a statistical power of 90% (1-β), we have to include 25 patients in each group.

>Sample size calculation based on data from stable CAD-patients on-aspirin<

The primary outcome is the difference in platelet aggregation between HTx patients with and without CAV and patients with stable CAD. From a previous study we know that the mean platelet aggregation in patients with stable coronary artery disease receiving aspirin is 324 aggregation units x minute with a standard deviation of 80 aggregation units x minute using AA as agonist (ASPI-test). Choosing a minimal relevant difference of 70 aggregation units x minute, a significance level (two-sided alpha) of 5%, and a statistical power of 90% (1-β), we have to include 28 patients in each group.

STATISTICS

Patients are divided into three groups according to the severity of CAV assessed by OCT (0%, 0-7% og >7% complex layered plaques). Platelet function are compared between groups. Normally distributed variables will be presented as mean ± SD. Non-parametric statistics and appropriate log-transformation will be performed if assumption of normality is not met. Between-group difference will be tested by Analysis of variance (ANOVA) or Kruskal-Wallis equality-of-populations rank test when appropriate. A two-tailed p-value of <0.05 or less will be considered statistically significant. Platelet variables in HTx patients before and after aspirin are compared to the same variables measured in healthy controls and stable CAD patients. Between-group difference will be tested by students t-test or Wilcoxon-Mann-Whitney test when appropriate.

PERSPECTIVES By combining advanced analyses and expert knowledge from the Department of Cardiology and the research unit at Department of Biochemistry, new knowledge regarding platelet function and ECP treatment in HTx patients will be obtained. Potentially, ECP treatments and medical therapy inhibiting platelets may reduce the development of CAV thus improving quality of life and long-term prognosis for HTx patients worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100
* Informed and signed consent
* Positive Luminex analysis: Blood samples with DSA levels >3000 MFI
* Coronary angiography with evidence of CAV (ISHLT class ≥1) according to ISHLT criteria's.

Exclusion Criteria:

* Severe asthma or COLD with FEV1 < 50%*
* 2° or 3° AV block*
* Pregnancy
* Creatinine >250 mmol/l**
* Platelet count below 20 x 109/L
* History of allergy to 8-Methoxypsoralen (8-MOP)
* History of light-sensitive disease

  * These patients will not be subjected to adenosine submission **These patients will not be subjected to OCT evaluation

Control groups:

* 120 patients with angiographically proven coronary artery disease treated with 75 mg aspirin daily for at least seven days (no other antithrombotic drugs are allowed). These data is already available.
* 60 healthy subjects on no medication - samples are taken before and after 75 mg aspirin daily for at least seven days. These data is already available.

As the data regarding the control groups are already available from previous studies at our department, these control patients are no considered actively included in this study. Hence, the patient population consists of the 60 HTx patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-10-13 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in CAV | Baseline and 12 months follow up
  Changes in CAV assessed by CAG, OCT and advanced echocardiography

SECONDARY OUTCOMES:
Platelet aggregation assessment related to CAV. | Baseline and 7 days after aspirin treatment.
  Platelet aggregation compared to healthy controls and patients with coronary artery disease.
Changes in platelet aggregation | Baseline and 7 days after aspirin treatment.
  Changes in platelet aggregation before and after aspirin
Changes in DSA levels | Baseline and 12 months follow up
  Changes in DSA levels before and after ECP-treatment
Changes in exercise and longitudinal myocardial deformation capacity | Baseline and 12 months follow up
  changes in exercise and longitudinal myocardial deformation capacity before and after ECP treatment.
Changes in CFVR | Baseline and 12 months follow up
  Changes in microvascular function assessed by CFVR before and after ECP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Eiskjær, Professor, Principal Investigator — Aarhus Universitetshospital, Afdeling for Hjertesygdomme, Palle Juul Jensens Blvd. 99, 8200 Aarhus N
Locations (1):
- Aarhus Universitetshospital, Afdeling for Hjertesygdomme, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clemmensen TS, Munk K, Tram EM, Ilkjaer LB, Severinsen IK, Eiskjaer H. Twenty years' experience at the Heart Transplant Center, Aarhus University Hospital, Skejby, Denmark. Scand Cardiovasc J. 2013 Dec;47(6):322-8. doi: 10.3109/14017431.2013.845688. Epub 2013 Oct 16. PMID 24131212
- [Background] Stehlik J, Edwards LB, Kucheryavaya AY, Benden C, Christie JD, Dipchand AI, Dobbels F, Kirk R, Rahmel AO, Hertz MI; International Society of Heart and Lung Transplantation. The Registry of the International Society for Heart and Lung Transplantation: 29th official adult heart transplant report--2012. J Heart Lung Transplant. 2012 Oct;31(10):1052-64. doi: 10.1016/j.healun.2012.08.002. No abstract available. PMID 22975095
- [Background] Berry GJ, Burke MM, Andersen C, Bruneval P, Fedrigo M, Fishbein MC, Goddard M, Hammond EH, Leone O, Marboe C, Miller D, Neil D, Rassl D, Revelo MP, Rice A, Rene Rodriguez E, Stewart S, Tan CD, Winters GL, West L, Mehra MR, Angelini A. The 2013 International Society for Heart and Lung Transplantation Working Formulation for the standardization of nomenclature in the pathologic diagnosis of antibody-mediated rejection in heart transplantation. J Heart Lung Transplant. 2013 Dec;32(12):1147-62. doi: 10.1016/j.healun.2013.08.011. PMID 24263017
- [Background] Patel J, Klapper E, Shafi H, Kobashigawa JA. Extracorporeal photopheresis in heart transplant rejection. Transfus Apher Sci. 2015 Apr;52(2):167-70. doi: 10.1016/j.transci.2015.02.004. Epub 2015 Feb 11. PMID 25748232
- [Background] Barten MJ, Dieterlen MT. Extracorporeal photopheresis after heart transplantation. Immunotherapy. 2014;6(8):927-44. doi: 10.2217/imt.14.69. PMID 25313571
- [Background] Matsuo Y, Cassar A, Li J, Flammer AJ, Choi BJ, Herrmann J, Gulati R, Lennon RJ, Kang SJ, Maehara A, Kitabata H, Akasaka T, Lerman LO, Kushwaha SS, Lerman A. Repeated episodes of thrombosis as a potential mechanism of plaque progression in cardiac allograft vasculopathy. Eur Heart J. 2013 Oct;34(37):2905-15. doi: 10.1093/eurheartj/eht209. Epub 2013 Jun 19. PMID 23782648
- [Background] Cassar A, Matsuo Y, Herrmann J, Li J, Lennon RJ, Gulati R, Lerman LO, Kushwaha SS, Lerman A. Coronary atherosclerosis with vulnerable plaque and complicated lesions in transplant recipients: new insight into cardiac allograft vasculopathy by optical coherence tomography. Eur Heart J. 2013 Sep;34(33):2610-7. doi: 10.1093/eurheartj/eht236. Epub 2013 Jun 25. PMID 23801824
- [Background] Arbustini E, Dal Bello B, Morbini P, Gavazzi A, Specchia G, Vigano M. Multiple coronary thrombosis and allograft vascular disease. Transplant Proc. 1998 Aug;30(5):1922-4. doi: 10.1016/s0041-1345(98)00526-0. No abstract available. PMID 9723334
- [Background] Modjeski KL, Morrell CN. Small cells, big effects: the role of platelets in transplant vasculopathy. J Thromb Thrombolysis. 2014 Jan;37(1):17-23. doi: 10.1007/s11239-013-0999-4. PMID 24264961
- [Background] Maeda A. Extracorporeal photochemotherapy. J Dermatol Sci. 2009 Jun;54(3):150-6. doi: 10.1016/j.jdermsci.2009.03.002. Epub 2009 Apr 14. PMID 19369039
- [Background] Ward DM. Extracorporeal photopheresis: how, when, and why. J Clin Apher. 2011;26(5):276-85. doi: 10.1002/jca.20300. Epub 2011 Sep 5. PMID 21898572
- [Background] Lu WH, Palatnik K, Fishbein GA, Lai C, Levi DS, Perens G, Alejos J, Kobashigawa J, Fishbein MC. Diverse morphologic manifestations of cardiac allograft vasculopathy: a pathologic study of 64 allograft hearts. J Heart Lung Transplant. 2011 Sep;30(9):1044-50. doi: 10.1016/j.healun.2011.04.008. Epub 2011 Jun 2. PMID 21640617
- [Background] Gould KL, Lipscomb K. Effects of coronary stenoses on coronary flow reserve and resistance. Am J Cardiol. 1974 Jul;34(1):48-55. doi: 10.1016/0002-9149(74)90092-7. No abstract available. PMID 4835753